CLINICAL TRIAL: NCT03507790
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Study to Evaluate the Safety and Efficacy of CT1812 in Subjects With Mild to Moderate Alzheimer's Disease.
Brief Title: A Study to Evaluate the Safety and Efficacy of CT1812 in Subjects With Mild to Moderate Alzheimer's Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COG0201; R01AG058660 (NIH); 2022-002326-27 (EudraCT Number)
Record Dates: First submitted 2018-04-10; First posted 2018-04-25 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Mild to Moderate Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Drug Evaluation

STUDY DESIGN:
Intervention Model Description: This is a multi-center Phase 2, randomized, double-blind, placebo-controlled, parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Treatment- CT1812 100 mg (Active Comparator): CT1812 at a dose of 100 mg
  Interventions: Drug: CT1812
- Active Treatment- CT1812 300 mg (Active Comparator): CT1812 at a dose of 300mg
  Interventions: Drug: CT1812
- Placebo Comparator - Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT1812 — Active Study Drug
  Other Names: Study Drug; zervimesine
  Arms: Active Treatment- CT1812 100 mg; Active Treatment- CT1812 300 mg
Drug: Placebo — Non-active study drug
  Other Names: Matching Placebo
  Arms: Placebo Comparator - Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel group 36 week multicenter Phase 2 study of two doses of CT1812 in adults with mild to moderate Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel group 36 week multicenter Phase 2 study of two doses of CT1812 in adults with mild to moderate Alzheimer's Disease (AD).

This Phase 2 study is designed to evaluate the safety of two doses of CT1812 administered once daily for 6 months in adults aged 50 to 85 who have been diagnosed with mild to moderate Alzheimer's disease. Randomized participants will receive 100 mg of CT1812, 300 mg of CT1812, or placebo once daily for 182 days. Exploratory endpoints that evaluate the effect of CT1812 on biomarkers are also included.

ELIGIBILITY:
Inclusion Criteria:

1. Men, and women of non-childbearing potential, 50-85 years of age inclusively, with a diagnosis of mild to moderate Alzheimer's disease according to the 2011 NIA-AA criteria and at least a 6 month decline in cognitive function documented in the medical record.

   i) Non-childbearing potential for women is defined as postmenopausal (last natural menses greater than 24 months) or undergone a documented bilateral tubal ligation or hysterectomy. If last natural menses less than 24 months, a serum FSH value confirming post-menopausal status can be employed.

   ii) Male participants who are sexually active with a woman of child-bearing potential must agree to use condoms during the trial and for 3 months after last dose unless the woman is using an acceptable means of birth control. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of: intrauterine device (IUD), male or female condom, diaphragm, sponge, and cervical cap.
2. Diagnostic confirmation by amyloid PET with florbetaben or another approved amyloid PET ligand. Previous amyloid imaging study with a positive result will be accepted. If none is available, then amyloid PET will be conducted during screening. Diagnostic confirmation by a CSF sample collected at the screening visit lumbar puncture in place of amyloid PET will also be acceptable
3. Neuroimaging (MRI) obtained during screening consistent with the clinical diagnosis of Alzheimer's disease and without findings of significant exclusionary abnormalities (see exclusion criteria, number 4). An historical MRI, up to 1 year prior to screening, may be used as long as there is no history of intervening neurologic disease or clinical events (such as a stroke, head trauma etc.) and the subject is without clinical symptoms or signs suggestive of such intervening events.).
4. MMSE 18-26 inclusive.

Exclusion Criteria:

1. Screening MRI (or historical MRI, if applicable) of the brain indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct >1 cm3, >3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (e.g. abscess or brain tumor such as meningioma). If a small incidental meningioma is observed, the medical monitor may be contacted to discuss eligibility..
2. Clinical or laboratory findings consistent with:

   1. Other primary degenerative dementia, (dementia with Lewy bodies, fronto-temporal dementia, Huntington's disease, Creutzfeldt-Jakob Disease, Down syndrome, etc.).
   2. Other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.).
   3. Seizure disorder.
   4. Other infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, other laboratory values etc.).
3. A current DSM-V diagnosis of active major depression, schizophrenia or bipolar disorder. Subjects with depressive symptoms successfully managed by a stable dose of an antidepressant are allowed entry.
4. Clinically significant, advanced or unstable disease that may interfere with outcome evaluations.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Caggiano, MD, Study Director — Cognition Therapeutics
Locations (32):
- United States (12):
  - 21st Century Neurology/ Xenoscience Inc., Phoenix, Arizona
  - Imaging Endpoints, Scottsdale, Arizona
  - Ki Health Partners, LLC dba New England Institute for Clinical Research, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Charter Research, Lady Lake, Florida
  - ClinCloud, LLC, Maitland, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Compass Research LLC- Bioclinica Research, The Villages, Florida
  - ClinCloud, Viera, Florida
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - The Ohio State University - Wexner, Columbus, Ohio
  - Neuro Behavirol Clinical Research C, North Canton, Ohio
- Australia (4):
  - St Vincent's Hospital Sydney, Ivanhoe, Victoria
  - Alfred Health, Melbourne, Victoria
  - Melbourne Health, Parkville, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Czechia (8):
  - Neuro Health Centrum ltd, Brno
  - NeuropsychiatrieHK S.R.O, Hradec Králové
  - A-Shine S.R.O, Pilsen
  - Clintrial S.R.O, Prague
  - Neuropsychiatrie s.r.o., Prague
  - Forbeli S.R.O, Prague
  - INEP, Prague
  - Vestra Clinics, Rychnov nad Kněžnou
- Netherlands (3):
  - Brain Research Den Bosch, 's-Hertogenbosch
  - Brain Research Center Amsterdam, Amsterdam
  - Brain Research Center Zwolle, Zwolle
- Spain (5):
  - Fundación ACE, Barcelona
  - Hospital Clinico Universitario Virgen De La Arrixaca, El Palmar
  - Centro de Salud San Juan, Salamanca
  - Hospital Victoria EUGENIA. Unidad de Neurociencias., Seville
  - Fundación Neuropolis - Hospital Viamed Montecanal, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lizama BN, North HA, Pandey K, Williams C, Duong D, Cho E, Di Caro V, Ping L, Blennow K, Zetterberg H, Lah J, Levey AI, Grundman M, Caggiano AO, Seyfried NT, Hamby ME. An interim exploratory proteomics biomarker analysis of a phase 2 clinical trial to assess the impact of CT1812 in Alzheimer's disease. Neurobiol Dis. 2024 Sep;199:106575. doi: 10.1016/j.nbd.2024.106575. Epub 2024 Jun 22. PMID 38914170
- See also: Shine Study Information — https://cogrx.com/tag/shine/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 12 centers in the United States, 3 centers in Australia, 3 centers in the Netherlands, 8 centers in Czech Republic, and 4 centers in Spain.
Pre-assignment Details: A total of 372 participants were screened, and 153 were randomized: 51 to CT1812 100 mg, 51 to CT1812 300 mg, and 51 to placebo. Study drug was administered to all participants in the CT1812 groups (100%) and to 50 participants (98.0%) in the placebo group. One participant in the placebo arm was randomized in error and did not receive study drug after informing the site post-randomization and prior to dosing of a prohibited concomitant medication.
Groups:
- Active Treatment- CT1812 300 mg: CT1812 at a dose of 300 mg
  CT1812: Active Study Drug
Period: Overall Study
Arm/Group | Active Treatment- CT1812 100 mg | Active Treatment- CT1812 300 mg | Placebo Comparator - Placebo
Started | 51 | 51 | 51 (One participant in the placebo arm was randomized in error and did not receive study drug after informing the site post-randomization and prior to dosing of a prohibited concomitant medication.)
Completed | 47 | 35 | 46
Not Completed | 4 | 16 | 5
Not completed — Adverse Event | 0 | 11 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Subject moved to another location | 1 | 2 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — COVID 19 Pandemic | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Discontinuation of the trial at the site | 1 | 1 | 0
Not completed — Randomized in error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the placebo arm was randomized in error and did not receive the study drug after informing the site, post-randomization and prior to dosing, about a prohibited concomitant medication. Therefore, the number of participants in the placebo arm is 50, not 51.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment- CT1812 100 mg | Active Treatment- CT1812 300 mg | Placebo Comparator - Placebo | Total
Number analyzed (Participants) | 51 | 51 | 50 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] — Data are based on the safety population, which is defined as all participants who received one or more doses of the study drug.
  years | 72.4 (6.96) | 74.1 (7.14) | 71.6 (7.97) | 72.7 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants] — Data are based on the safety population, which is defined as all participants who received one or more doses of the study drug.
  Participants
    Female | 34 | 29 | 28 | 91
    Male | 17 | 22 | 22 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data are based on the safety population, which is defined as all participants who received one or more doses of the study drug.
  Participants
    Hispanic or Latino | 4 | 6 | 1 | 11
    Not Hispanic or Latino | 47 | 44 | 49 | 140
    Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data are based on the safety population, which is defined as all participants who received one or more doses of the study drug.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
    Black or African American | 0 | 1 | 2 | 3
    White | 50 | 49 | 47 | 146
    More than one race | 0 | 1 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] — Data are based on the safety population, which is defined as all participants who received one or more doses of the study drug. Population: Two subjects-one in the CT1812 100 mg arm and one in the CT1812 300 mg arm-missed the baseline height measurement.
  cm
    number analyzed (Participants) | 50 | 50 | 50 | 150
    (all) | 165.77 (9.143) | 165.88 (11.802) | 167.52 (9.998) | 166.39 (10.335)
Weight [Mean (Standard Deviation); unit: Kg] — Data are based on the safety population, which is defined as all participants who received one or more doses of the study drug.
  Kg | 72.01 (15.105) | 67.85 (13.268) | 68.10 (12.672) | 69.33 (13.770)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Data are based on the safety population, which is defined as all participants who received one or more doses of the study drug. Population: Two subjects-one in the CT1812 100 mg arm and one in the CT1812 300 mg arm-missed the baseline BMI measurement.
  kg/m^2
    number analyzed (Participants) | 50 | 50 | 50 | 150
    (all) | 26.04 (4.574) | 24.43 (3.554) | 24.13 (3.046) | 24.87 (3.846)

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants With at Least One Mild, Moderate, or Severe Treatment Emergent Adverse Events (TEAEs)
Description: Adverse events were captured from the start of study-related procedures at Visit 1 (including diagnostic assessments or signing of ICF) onward during the course of this study. Adverse events were coded using MedDRA Version 27.0.TEAEs are events that occurred or worsened on or after the first application of study drug. Participants are counted once for each system organ class (SOC) and once for each preferred term (PT).
Time Frame: Up to 210 Days
Population: Data are based on the safety population, which is defined as all participants who received one or more doses of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment- CT1812 100 mg | Active Treatment- CT1812 300 mg | Placebo Comparator - Placebo
Number analyzed (Participants) | 51 | 51 | 50
Participants
  All TEAEs | 36 | 42 | 39
  Mild TEAEs | 19 | 22 | 22
  Moderate TEAEs | 16 | 16 | 14
  Severe TEAEs | 1 | 4 | 3

2. Primary Outcome: Number of Study Participants With at Least One Treatment Emergent Adverse Events (TEAs) and Serious Adverse Events (SAEs).
Description: as for outcome 1
Time Frame: Up to 210 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment- CT1812 100 mg | Active Treatment- CT1812 300 mg | Placebo Comparator - Placebo
Number analyzed (Participants) | 51 | 51 | 50
Participants
  Participants with at least one TEAE | 36 | 42 | 39
  Participants with at least one TEAE related to treatment | 11 | 16 | 7
  Participants with a TEAE leading to study drug discontinuation | 0 | 11 | 3
  Participants with a TEAE leading to death | 0 | 0 | 1
  Participants with at least one SAE | 2 | 3 | 5
  Participants with at least one SAE related to treatment | 0 | 1 | 0

3. Secondary Outcome: Change From Baseline in the Cerebrospinal Fluid (CSF) Biomarkers
Description: Change from baseline in CSF-Aβ, Tau, phospho-Tau, neurogranin, synaptotagmin, synaptosomal-associated protein-25 (SNAP25), neurofilament light chain (NfL), and Aβ-oligomers.Change from baseline is calculated as the observed value minus the baseline value.
Time Frame: Baseline to Day 182
Population: The analyzed population represents the number of subjects in the Efficacy modified intent-to-treat (mITT) population and participants who had both baseline and Day 182 CSF samples collected.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Active Treatment- CT1812 100 mg | Active Treatment- CT1812 300 mg | Placebo Comparator - Placebo
Number analyzed (Participants) | 51 | 50 | 49
ng/L
  Alpha Synuclein Protein (ASYNP) (ng/L) - Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 17 | 10 | 16
  Alpha Synuclein Protein (ASYNP) (ng/L) - Concentration change in CSF from Baseline to Day 182 | 48.6 (625.13) | 38.3 (213.10) | -831.2 (3056.97)
  Amyloid Beta 1-40 (Aβ40) (ng/L) -Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 23 | 18 | 24
  Amyloid Beta 1-40 (Aβ40) (ng/L) -Concentration change in CSF from Baseline to Day 182 | -573.9 (2228.80) | -1076.7 (1781.36) | -17.9 (1633.79)
  Amyloid Beta 1-42 (Aβ42) (ng/L) -Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 23 | 18 | 24
  Amyloid Beta 1-42 (Aβ42) (ng/L) -Concentration change in CSF from Baseline to Day 182 | -13.5 (105.66) | -72.1 (121.62) | 3.1 (90.90)
  Glial Fibrillary Acidic Protein (GFAP) (ng/L) - Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 19 | 11 | 17
  Glial Fibrillary Acidic Protein (GFAP) (ng/L) - Concentration change in CSF from Baseline to Day 182 | -81.9 (457.85) | -87.4 (176.01) | -69.1 (321.21)
  Neurofilament Light Chain Protein (NFLP) (ng/L) Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 24 | 17 | 24
  Neurofilament Light Chain Protein (NFLP) (ng/L) Concentration change in CSF from Baseline to Day 182 | 72.8 (317.59) | -55.5 (262.24) | 297.7 (535.60)
  Neurogranin (NRGR) (ng/L) - Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 24 | 18 | 24
  Neurogranin (NRGR) (ng/L) - Concentration change in CSF from Baseline to Day 182 | 19.70 (82.557) | -22.77 (68.348) | -16.93 (44.348)
  Phosphorylated Tau Protein 181 (pTau181) (ng/L) Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 24 | 18 | 24
  Phosphorylated Tau Protein 181 (pTau181) (ng/L) Concentration change in CSF from Baseline to Day 182 | -0.74 (37.227) | -9.76 (45.506) | -4.03 (13.185)
  Synaptosomal-Associated Protein 25 (SNAP25) Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 24 | 17 | 24
  Synaptosomal-Associated Protein 25 (SNAP25) Concentration change in CSF from Baseline to Day 182 | -0.88 (6.485) | -1.64 (4.767) | -1.04 (3.763)
  Synaptotagmin (SYN) Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 24 | 17 | 24
  Synaptotagmin (SYN) Concentration change in CSF from Baseline to Day 182 | 0.75 (15.041) | -19.44 (98.693) | 4.66 (56.365)
  Tau Protein (TPROT) (ng/L) Concentration change in CSF from Baseline to Day 182: number analyzed (Participants) | 24 | 18 | 24
  Tau Protein (TPROT) (ng/L) Concentration change in CSF from Baseline to Day 182 | -8.4 (204.92) | -47.8 (358.68) | -9.4 (80.67)

4. Secondary Outcome: Amyloid Beta 1-42/Amyloid Beta 1-40 (Aβ42/40) in the Cerebrospinal Fluid (CSF) Biomarkers
Description: Ratio of Amyloid Beta 1-42 (Aβ42) to Amyloid Beta 1-40 (Aβ40) Concentration from Baseline to Day 182.
Time Frame: Baseline to Day 182
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Active Treatment- CT1812 100 mg | Active Treatment- CT1812 300 mg | Placebo Comparator - Placebo
Number analyzed (Participants) | 51 | 50 | 49
ratio | 0.019 (0.0766) | -0.024 (0.0631) | -0.002 (0.0594)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the start of study-related procedures at Visit 1 (- 60 to -1 days) until the safety follow up visit V15 (study day 210 (±2) days). Important medical events and conditions occurring prior to this period were not recorded as AEs; they were captured within the medical chart and in the medical history section of the CRF.
Description: The safety of CT1812 was evaluated by the incidence and severity of adverse events (AEs) and changes in the usage of concomitant medications, vital signs, physical examination findings, electrocardiogram (ECG) findings, clinical laboratory testing (serum chemistry, hematology, and urinalysis), and Columbia-Suicide Severity Rating Scale (C-SSRS).
Arm/Group | Active Treatment- CT1812 100 mg | Active Treatment- CT1812 300 mg | Placebo Comparator - Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 1/50
Serious Adverse Events (participants affected / at risk) | 2/51 | 3/51 | 5/50
Other Adverse Events (participants affected / at risk) | 25/51 | 25/51 | 33/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment- CT1812 100 mg (N=51) | Active Treatment- CT1812 300 mg (N=51) | Placebo Comparator - Placebo (N=50)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infection unknown etiology (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Recurrent Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope x2 (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (intermittent) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Oncocytosis (left kidney) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Papillary Renal Cell Carcinoma (left kidney) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Retinal Detachment Right Side (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Lung Neoplasia Inferior Right with Metastasis in Liver and Bones (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment- CT1812 100 mg (N=51) | Active Treatment- CT1812 300 mg (N=51) | Placebo Comparator - Placebo (N=50)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 8 (8) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 7 (10) | 2 (2) | 4 (5)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 4 (4)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 4 (5)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 7 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2)
Blood potassium increased (Investigations) | 0 (0) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT03507790/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03507790/SAP_001.pdf